CLINICAL TRIAL: NCT04491682
Title: Megestrol Acetate Plus Rosuvastatin in Young Women With Atypical Endometrial Hyperplasia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Principle investigator, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53211029-01
Record Dates: First submitted 2020-06-21; First posted 2020-07-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Atypical Endometrial Hyperplasia
Keywords: megestrol acetate; rosuvastatin; atypical endometrial hyperplasia; conservative treatment
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Megestrol Acetate; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MA + Rosuvastatin (Experimental): Patients will receive MA 160 mg and rosuvastatin 10 mg by mouth daily for at least 6 months.Then every 3 months, hysteroscopy will be used to evaluate the endometrial condition, and findings will be recorded.
  Due to personal reasons, it may not be possible to accept hysteroscopic evaluation every three months, then the longest duration will be 8 months.
  Interventions: Drug: Megestrol Acetate; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Megestrol Acetate — At a dosage of 160 mg/day
Drug: Rosuvastatin — At a dosage of 10 mg/day

SUMMARY:
To see if megestrol acetate plus rosuvastatin will be superior to reversing the endometrial lesion to a normal endometrium than megestrol acetate alone in patients with atypical endometrial hyperplasia (AEH). Considering the large sample size in RCT, we used Simon two-stage design.

DETAILED DESCRIPTION:
After diagnosed of AEH by hysteroscopy, patients will be enrolled. Age, height, weight, waist circumstances, blood pressure, basic history of infertility and blood pressure will be collected. Blood tests, including fasting blood glucose (FBG), fasting insulin (FINS), OGTT 2h blood glucose and insulin, blood lipids, SHBG, sex hormone levels, anti-müllerian hormone(AMH), creatine kinase(CK) and renal/liver function tests will be performed before treatment to evacuate their basic conditions. Each subject will receive body fat testing by Inbody 520.

Patients are randomized to 1 of 2 treatment groups. Patients will receive MA 160 mg plus rosuvastatin 10mg by mouth daily for at least 6 months. Then hysteroscopy will be used to evaluate the endometrial condition every 3 months, and intra-operative findings will be recorded. Complete response (CR) is defined as the reversion of endometrial atypical hyperplasia to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia without atypic; stable disease (SD) is defined as the persistence of the disease; and progressive disease (PD) is defined as the appearance of endometrial cancer in patients. Continuous therapies will be needed in PR or NR. Patients with PD will be recommended for hysterectomy.

Two months of maintenance treatment will be recommended for patients with CR, and participants will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed pathological diagnosis based upon hysteroscopy
* Have a desire for remaining reproductive function or uterus
* Good compliance with adjunctive treatment and follow-up
* Abnormal blood lipid. At least meet one of the following five items:

  1. Total cholesterol (TC) ≥ 5.2mmol/L (200mg/dL)
  2. Low-density lipoprotein cholesterol (LDL-C) ≥ 3.4mmol/L (130mg/dL)
  3. Fasting triglycerides (TG) ≥ 1.7mmol/L (150mg/dL)
  4. High-density lipoprotein cholesterol (HDL-C) < 1.03mmol/L (40mg/dL)
  5. Apo-lipoprotein-A (Apo-A) < 1.0g/L

Exclusion Criteria:

* Acute liver disease or liver tumor (benign or malignant) or renal dysfunction
* Pregnancy or potential pregnancy
* Under treatment of high-dose progestin therapy more than 1 months in recent 6 months
* Confirmed diagnosis of any cancer in reproductive system
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Hypersensitivity or contradiction for using MA or statins
* Already diagnosed with hyperlipidemia and using lipid-lowering drugs
* With other factors of reproductive dysfunction;
* Strong request for uterine removal or other conservative treatment
* Smoker (>15 cigarettes a day)
* Drinker (>20 grams a day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Pathological response rate | 12 to 16 weeks
  From date of randomization or initial therapy until the date of CR or date of hysterectomy, whichever come first, assessed up to 16 weeks.

SECONDARY OUTCOMES:
Pathological response rate | 28 to 32 weeks
  From date of randomization or initial therapy until the date of CR or date of hysterectomy, whichever come first, assessed up to 32 weeks.
Pathological response duration | Up to 2 years
  Pathological response duration
Pathological response rate classified by different blood lipid level | Up to 32 weeks
  Pathological response rate classified by different blood lipid level
Toxicity evaluation | Up to 32 weeks
  Toxicity evaluation according to CTCAE 5.0 version.
Relapse rate | up to 2 years after the therapy for each patient
Pregnancy rate | up to 2 years after the therapy for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Chen, Principal Investigator — Obstetrics and Gynecology Hospital, Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, China